CLINICAL TRIAL: NCT00742677
Title: Early Oral Feeding After a Gynaecologic Oncologic Laparotomy: A Randomized Controlled Trial
Brief Title: Feeding Schedules After Surgery in Patients With Gynecologic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000612328; IEO-S328/506
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-07

CONDITIONS: Female Reproductive Cancer
Keywords: female reproductive cancer
MeSH Terms: interventions — Nutritional Support

ARMS (2):
- Group 1 (early feeding) (Experimental): Patients are offered a liquid diet on day 1 for 24 hours following surgery. Beginning on day 2, patients who tolerate a liquid diet are offered a light regular diet until hospital discharge.
  Interventions: Procedure: nutritional support
- Group 2 (traditional feeding) (Active Comparator): Patients are offered nothing by mouth on days 1 and 2 following surgery. Beginning on day 3, patients are offered a liquid diet for 24 hours. Beginning on day 4, patients who tolerate a liquid diet (absence of nausea and vomiting) are offered a semi-solid diet for 24 hours. Beginning on day 5, patients who tolerate a semi-solid diet are offered a light regular diet until hospital discharge.
  Interventions: Procedure: nutritional support

INTERVENTIONS:
Procedure: nutritional support — Given orally

SUMMARY:
RATIONALE: Abdominal pain and nausea and vomiting may be lessened by waiting after surgery before eating foods by mouth. It is not yet known which feeding schedule is more effective in patients undergoing surgery.

PURPOSE: This randomized clinical trial is comparing two feeding schedules after laparotomy in patients with gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the relationship between the different policies of realimentation (early oral feedings versus traditional feedings) and the length of hospital stay following a laparotomy in patients with gynecologic oncologic disease.
* To assess the degree of postoperative abdominal pain in these patients.
* To evaluate the incidence of ileus symptoms, including nausea and vomiting, and the postoperative recovery of intestinal activity in these patients.
* To determine the incidence of postoperative complications in these patients.
* To elucidate the global postoperative patient's satisfaction and the quality of life in both groups of patients.

OUTLINE: Patients are stratified according to laparotomy with or without intestinal resection (yes vs no), and presence of ovarian cancer (yes vs no). Patients are randomized to 1 of 2 groups at the end of surgery.

* Group 1 (early feeding): Patients are offered a liquid diet on day 1 for 24 hours following surgery. Beginning on day 2, patients who tolerate a liquid diet are offered a regular diet until hospital discharge.
* Group 2 (traditional feeding): Patients are offered nothing by mouth on days 1 and 2 following surgery. Beginning on day 3, patients are offered a liquid diet for 24 hours. Beginning on day 4, patients who tolerate a liquid diet (i.e., no nausea and vomiting) are offered a semi-solid diet for 24 hours. Beginning on day 5, patients who tolerate a semi-solid diet are offered a light regular diet until hospital discharge.

Data is collected through the Post-Operative Pain Questionnaire, Bowel Function Table, Global Postoperative Patient's Satisfaction Questionnaire, Postoperative Complication and Hospital Stay Questionnaire, and the Quality of Life Questionnaires EORTC OV-28 and EORTC QLQ-C30.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Preoperative diagnosis for probable gynecologic pathology

  * No benign pathology or final histopathology diagnosis confirmed as non-gynecologic disease
* Admitted to the European Institute of Oncology
* Elected to undergo laparotomic surgery

  * No total or anterior pelvic exenteration
  * No emergency laparotomy

PATIENT CHARACTERISTICS:

* No metabolic pathology (e.g., diabetes mellitus type I)
* No preoperative ASA score ≥ 4
* No preoperative infection
* No severe malnutrition (weight loss > 10% within the past 3 months)
* No preoperative intestinal obstruction
* No postoperative admission to the intensive care unit (ICU) for more than 24 hours
* No severe concomitant medical condition

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior abdominal and/or pelvis radiotherapy

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay

SECONDARY OUTCOMES:
Incidence of symptoms of postoperative ileus (e.g., nausea, vomiting, time to feel intestinal activity, time to passage of flatus, and time to bowel movement)
Degree of postoperative abdominal pain
Global postoperative patient satisfaction
Quality of life using the EORTC OV-28 and EORTC QLQ-C30 questionnaires at baseline and at day 30
Postoperative requirement of antiemetic and analgesic medication
Postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Minig, MD, Principal Investigator — European Institute of Oncology; Roberto Biffi, MD, Principal Investigator — European Institute of Oncology; Angelo Maggioni, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy